CLINICAL TRIAL: NCT06696755
Title: A Phase 2, Multicenter, 6-Week, Double Blind, Placebo- Controlled Study to Evaluate the Efficacy and Safety of Icalcaprant in Subjects With Bipolar Depression
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Oral Icalcaprant in Adult Participants With Bipolar I or II Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M25-526
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Bipolar I Disorder; Bipolar II Disorder
Keywords: Bipolar I Disorder; Bipolar II Disorder; Bipolar Disorder; lcalcaprant; ABBV-1354; CVL-354
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Icalcaprant Dose A (Experimental): Participants will receive oral Icalcaprant dose A once daily for 6 weeks and followed for 4 weeks.
  Interventions: Drug: Icalcaprant
- Group 2: Icalcaprant Dose B (Experimental): Participants will receive oral Icalcaprant dose B once daily for 6 weeks and followed for 4 weeks.
  Interventions: Drug: Icalcaprant
- Group 3: Placebo for Icalcaprant (Placebo Comparator): Participants will receive oral placebo for Icalcaprant daily for 6 weeks and followed for 4 weeks.
  Interventions: Drug: Placebo for Icalcaprant

INTERVENTIONS:
Drug: Icalcaprant — Oral Capsules
  Other Names: ABBV-1354; CVL-354
  Arms: Group 1: Icalcaprant Dose A; Group 2: Icalcaprant Dose B
Drug: Placebo for Icalcaprant — Oral Capsules
  Arms: Group 3: Placebo for Icalcaprant

SUMMARY:
Bipolar disorder is a severe chronic mood disorder that affects up to 4% of the adult population and 1.8% of the pediatric population in the United States. This study will assess how safe and effective Icalcaprant is in treating adult participants with bipolar I or II disorder.

Icalcaprant is an investigational drug being developed for the treatment of depressive episodes in adult participants with bipolar I or II disorder. Participants are placed in 1 of 3 groups, called treatment arms. There is a 1 in 3 chance that a participant will be assigned to a placebo. Around 195 adult participants with bipolar I or II disorder will be enrolled in approximately 35 sites across the United States of America.

Participants will receive oral capsules of Icalcaprant or matching placebo once daily for 6 weeks, with a 4-week safety follow-up period.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of bipolar I or II according to the (Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) DSM-5-TR) without psychotic features, confirmed by the Mini International Neuropsychiatric Interview (MINI) 7.0.2, and currently experiencing an (major depressive episode) MDE beginning at least 4 weeks prior to consent and not exceeding 6 months prior to screening.
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 35.0 kg/m^2.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.
* CGI-S-BP score of ≥ 4 for depression and overall bipolar illness at screening (Visit 1) and baseline (Visit 2).
* YMRS total score ≤ 12 at screening (Visit 1) and baseline (Visit 2).
* Participants on treatment with a single mood stabilizer (lithium, valproate, or lamotrigine), maintained at a stable dose for ≥ 28 days prior to screening. Current mood stabilizer dose must remain unchanged for the duration of the study.

  * If taking lithium or valproate, participant must have a therapeutic blood level at screening of lithium (0.8 - 1.2 mg/dL) or valproate (50 - 125 mg/dL).
  * If taking lamotrigine, participant must be taking a locally approved maintenance dose.

Exclusion Criteria:

* History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.
* History of or active medical conditions(s) that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the subject's well-being. This includes any unstable condition, history or evidence of malignancy (other than treated basal or squamous cell carcinoma), or any significant hematologic, endocrine, cardiovascular, respiratory, renal, hepatic, gastrointestinal, or neurological disorder (if there is a history of such disease but the condition has been stable for more than 1 year, does not require treatment with prohibited medications, and is judged by the investigator not to interfere with the participant's participation in the study, the participant may be included in the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 6 in the MADRS (Montgomery-Åsberg Depression Rating Scale) total score | Up to approximately Week 6
  MADRS is a depression rating scale consisting of 10 items representing the core symptoms of depressive illness, each rated 0 (no symptom) to 6 (severe symptom). Total score ranges from 0 (no depression) to 60 (severely depressed).
Number of Participants with Adverse Events (AEs) | Up to approximately 10 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study

SECONDARY OUTCOMES:
Change from Baseline to Week 6 in Clinician Global Impression of Severity - Bipolar Disorder (CGI-S-BP) score | Up to approximately Week 6
  Clinician Global Impression of Severity - Bipolar Disorder (CGI-S-BP) is a clinician-reported measure of severity of mania, depression, and overall bipolar disorder. Clinicians are asked to consider their total clinical experience with bipolar subjects and assess how severely ill has the participant been during the past 7 days. Response options range from 'Normal, not ill' to 'Very severely ill'.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-526